CLINICAL TRIAL: NCT07252336
Title: A Multicenter Study of CD19 CAR-T Cells in the Treatment of Adult Patients With Primary Ph Chromosome Positive Acute Lymphoblastic Leukemia
Brief Title: A Multicenter Study of CAR-T Cells in Primary Ph+All
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Zhejiang University (Other)
Collaborators: Yake Biotechnology Ltd. (Industry)
Responsible Party: Principal Investigator, He Huang, Clinical Professor, Zhejiang University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TXB2025020
Record Dates: First submitted 2025-11-18; First posted 2025-11-26 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-11

CONDITIONS: ALL
Keywords: CD19 CAR-T

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CAR-T cells（ chimeric antigen receptor T cells） (Experimental): CD19 CAR-T 2×10e6 CAR+ T cells/kg,
  Interventions: Drug: CD19 CAR-T cells

INTERVENTIONS:
Drug: CD19 CAR-T cells — Each subject receive CD19/CD22 CAR T-cells by intravenous infusion

SUMMARY:
A Multicenter Study of CD19 CAR-T Cells in the Treatment of Adult Patients With Primary Ph Chromosome Positive Acute Lymphoblastic Leukemia

DETAILED DESCRIPTION:
This study is a single-arm, open-label, multicenter clinical trial that plans to enroll approximately 50 adult patients with newly diagnosed Ph-positive acute lymphoblastic leukemia to undergo CD19 CAR-T cell therapy. The primary objective is to evaluate the efficacy of CD19 CAR-T therapy in adult patients with newly diagnosed Ph-positive acute lymphoblastic leukemia. The secondary objective is to assess the safety of CD19 CAR-T therapy in this patient population. The exploratory objectives include evaluating the in vivo expansion and persistence of CAR-T cells, as well as B-cell depletion.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years old, gender not restricted;
2. Subjects diagnosed with B-cell acute lymphoblastic leukemia (B-ALL) in accordance with the 2016 WHO Classification of Acute Leukemias;
3. Abnormal B cells positive for CD19 and CD22 by immunophenotyping;
4. Subjects positive for Philadelphia chromosome (Ph chromosome) and BCR/ABL1 fusion gene by chromosomal and corresponding genetic testing;
5. Newly diagnosed B-ALL patients who have not received treatment with standard chemotherapy regimens;
6. Serum total bilirubin ≤ 51 μmol/L, serum ALT and AST both ≤ 3 times the upper limit of the normal reference range, and serum creatinine ≤ 176.8 μmol/L;
7. Left ventricular ejection fraction (LVEF) ≥ 50% as assessed by echocardiography;
8. Subjects with no active pulmonary infection and oxygen saturation ≥ 92% without oxygen supplementation;
9. Estimated survival time ≥ 3 months;
10. ECOG performance status score 0-2;
11. Females and males of childbearing potential must agree to use appropriate contraceptive measures before enrollment, during study participation, and within 6 months after infusion;
12. Subjects voluntarily participate in this study and sign the informed consent form.

Exclusion Criteria:

* Subjects meeting any of the following exclusion criteria are ineligible for enrollment in this study:

  1. Subjects with a history of epilepsy or other central nervous system diseases;
  2. Subjects with a prior history of QT interval prolongation or severe cardiac diseases;
  3. Pregnant or lactating women (the safety of this therapy for unborn children is unknown);
  4. Subjects with untreated active infections;
  5. Subjects with serological evidence of chronic hepatitis B virus (HBV) infection who are unable or unwilling to receive standard prophylactic antiviral treatment, or have a detectable HBV viral DNA load; subjects with serological evidence of hepatitis C virus (HCV) infection who have not completed curative treatment or have a detectable HCV viral load;
  6. Human immunodeficiency virus (HIV) antibody positive;
  7. Syphilis antibody positive;
  8. Subjects who have previously received any gene therapy products;
  9. Subjects with other uncontrolled diseases who, in the investigator's judgment, are unsuitable for enrollment;
  10. Any other conditions that, in the investigator's judgment, may increase the risk to the subject or interfere with the study results.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-11-30 (Estimated); Primary Completion 2027-11-30 (Estimated); Study Completion 2028-11-30 (Estimated)

PRIMARY OUTCOMES:
Complete Molecular Response Rate after CD19 CAR-T Cell Therapy | 28 days after infusion
  Laboratory tests

SECONDARY OUTCOMES:
Leukemia-Free Survival | 2 years after infusion
  Survival follow-up
Overall survival | 2 years after infusion
  Survival follow-up
Cumulative Incidence of Relapse | 2 years after infusion
  Laboratory tests
Complete Molecular Response Rate after CD22 CAR-T Cell Therapy | 2 years after infusion
  Laboratory tests

CONTACTS AND LOCATIONS:
Locations (1):
- The first affiliated hospital of medical college of zhejiang university, Hangzhou, Zhejiang, China